CLINICAL TRIAL: NCT05664165
Title: Can the Efficiency of Dry Needling and Cold Spray-stretching Treatments be Documented by Ultrasonography and Electrophysiology?
Brief Title: The Efficiency of Dry Needling and Cold Spray-stretching Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Duygu Geler Külcü, Prof, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HNEAH-KAEK 2019/38
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Myofascial Pain Syndromes; Myofascial Trigger Point Pain
Keywords: cold spray; dry neddling; histogram; trigger point
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): It was performed using a deep dry needling technique using 0.25x25 mm disposable sterile steel acupuncture needles (HuaLong, China) while patient was in prone position. The needle inserted in the trigger point and stimulation was performed by manipulating it up and down several times. The needle was kept in the trigger point for 1-3 minutes and removed after the muscle spasm regressed . One session per week, a total of 3 sessions were applied.
  Interventions: Other: dry needling
- Cold spray and stretching (Experimental): The patient was placed on the chair with the head and body upright in the most comfortable position possible and voluntary relaxation was achieved. One end of the muscle was fixed in order to apply passive stretching. The cooler spray (in its content; 0.06% menthol, 2.06% isopropyl alcohol, 2% isopropyl alcohol) was sprayed to the surface at an angle of 30° from a distance of approximately 30-50 cm, while passive stretching was applied. One session per week, a total of 3 sessions were applied
  Interventions: Other: cold spray and stretching

INTERVENTIONS:
Other: dry needling — The needle inserted in the trigger point and stimulation was performed by manipulating it up and down several times. The needle was kept in the trigger point for 1-3 minutes and removed after the muscle spasm regressed
  Arms: Dry needling
Other: cold spray and stretching — The cooler spray (in its content; 0.06% menthol, 2.06% isopropyl alcohol, 2% isopropyl alcohol) was sprayed to the surface at an angle of 30° from a distance of approximately 30-50 cm, while passive stretching was applied.
  Arms: Cold spray and stretching

SUMMARY:
A prospective randomized single-blind study included 60 patients aged 18-65 years who have MPS with active triger points in the upper trapezius muscle. Patients were randomized into two treatment groups as dry needling (DN) and cold spray-stretching. Both treatment groups received 1 treatment per week and totally 3 sessions. Evaluation parameters were pain level assessed by visual analog scale (VAS) and algometer, neck range of motion angles, functional level assessed by neck disability index (NDI). The effects of the treatments on active trigger points were evaluated by sEMG and US histogram. All parameters were evaluated at the beginning of the treatment and after 3 sessions of treatment. Algometer and sEMG were performed also before and after the 1st and 3rd sessions.

DETAILED DESCRIPTION:
OBJECTIVE: To compare the efficacy of dry needling and cold spray stretching treatments using surface electromyography (sEMG) and ultrasound (US) in the treatment of patients with myofascial pain syndrome (MPS) with active trigger point (TrP) in the upper trapezius muscle.

MATERIAL AND METHODS: A prospective randomized single-blind study included 60 patients aged 18-65 years who have MPS with ATP in the upper trapezius muscle. Patients were randomized into two treatment groups as dry needling (DN) and cold spray-stretching. Both treatment groups received 1 treatment per week and totally 3 sessions. Evaluation parameters were pain level assessed by visual analog scale (VAS) and algometer, neck range of motion angles, functional level assessed by neck disability index (NDI). The effects of the treatments on aTP were evaluated by sEMG and US histogram. All parameters were evaluated at the beginning of the treatment and after 3 sessions of treatment. Algometer and sEMG were performed also before and after the 1st and 3rd sessions.

ELIGIBILITY:
Inclusion Criteria:

* neck and / or back pain for at least 3 months,
* pain level> 3 in VAS measurement
* presence of active trigger point in upper trapezius muscle

Exclusion Criteria:

* cervical radiculopathy
* history of neck and / or shoulder surgery
* dry needling treatment in the neck and / or shoulder area in the last 1 month
* coagulation disorder and / or use of anticoagulant therapy
* migraine or dementia
* pacemaker
* needle phobia
* allergies to the substances in the coolant spray to be used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
pain intensity1 | Change from baseline at 3rd week
  Visual Analog Scale: The Visual Analog Scale (VAS) (0-10 cm) was used to record each patient's current level of neck pain, with 0 indicating no pain and 10 indicating the worst pain that the patient had experienced.Higher scores mean worse outcome
cervical range of motion angles | Change from baseline at 3rd week
  measured by goniometer for flexion, extension, left and right lateral flexion of cervical spine
pain intensity2 | Change from baseline at 3rd week
  Algometer: The pain threshold was measured before and after the the first and third sessions with a pressure algometer (Electronic Algometer Commander-USA) in kg / cm². The applied pressure was increased until the point the patient first felt the pain. Measurements were repeated 3 times and the mean average score was recorded.
Disability level | Change from baseline at 3rd week
  Neck Pain Disability Scale: The questionnaire consists of 20 items and measures neck movements, pain intensity, effect of neck pain on emotion factors, and interference with daily life activities. Each section is scored on a 0-5 rating scale and total score ranges from 0 to 100. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Gray Scale Ultrasonography | Change from baseline at 3rd week
  The upper trapezius muscle, where the trigger point was located, is visualized with US, and the images containing the focal, hypoechoic area (trigger point) in the middle of the muscle are recorded. The echogenicity values of these images is analyzed with ImageJ software.
Surface electromyography | Change from baseline at 3rd week
  While the patient was sitting on a chair, EMG electrodes were placed in the middle of the upper trapezius muscle between the seventh cervical vertebra (C7) and the acromion, covering the trigger point area. The patient was asked to keep the trapezius muscle in the resting position for six seconds, the average of the recordings repeated 3 times with 1 minute intervals was evaluated as resting EMG activity. Then he was asked to raise both shoulders and hold this position in isometric contraction for six seconds. The maximum and average amplitude values obtained from the recordings that were repeated 3 times with 1 minute intervals were also averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Külcü, prof, Principal Investigator — Haydarpaşa Numune Edutation and Research Hospital
Locations (1):
- Haydarpaşa Numune Education and Research Hospital, Istanbul, Turkey (Türkiye)